CLINICAL TRIAL: NCT02166853
Title: Effect of Early 48-hour Sevoflurane Inhalation on Gas Exchange and Inflammation in Patients Presenting With Acute Respiratory Distress Syndrome (ARDS) : a Monocentric, Prospective, Randomized Study.
Brief Title: Effects of SEvoflurane on Gas Exchange and Inflammation in Patients With ARDS (SEGA Study)
Acronym: SEGA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0195; 2013-005389-21
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome (ARDS); Sevoflurane; Mechanical ventilation; Intensive Care Unit (ICU); Prospective study; Lung injury; Gas exchange; Inflammation; Receptor for advanced glycation end-produts (RAGE); sRAGE
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Injury; Inflammation | interventions — Sevoflurane; Midazolam

ARMS (2):
- conventional group (Experimental): a "conventional group", in which intravenous sedation with midazolam will be administered
  Interventions: Drug: midazolam
- sevoflurane group (Experimental): a "sevoflurane group", in which patients will inhale sevoflurane during a 48 hour-period, through dedicated devices
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: sevoflurane — Sedation with inhaled sevoflurane
  Arms: sevoflurane group
Drug: midazolam — Sedation with intravenous midazolam
  Arms: conventional group

SUMMARY:
Numerous trials support the efficacy and safety of volatile anesthetic agents, namely inhalation of sevoflurane through dedicated devices, for the sedation of ICU patients. Several preclinical studies have shown that sevoflurane inhalation improves gas exchange and decreases pulmonary and systemic inflammation in experimental models of acute respiratory distress syndrome (ARDS).

The purpose of our prospective monocentric, randomized, controlled trial is to evaluate the effects of an early 48-hour sevoflurane inhalation on gas exchange and inflammation in patients with ARDS.

DETAILED DESCRIPTION:
BACKGROUND:

Acute respiratory distress syndrome (ARDS) is characterized by hypoxemic respiratory failure that can be lethal in 30 to 60% of patients. Its pathophysiological landmark, diffuse alveolar damage, is associated with alveolar inflammation, epithelial injury and alveolar fluid clairance impairment.

Several preclinical studies have shown that early sevoflurane inhalation improves gas exchange, reduces alveolar edema and attenuates pulmonary and systemic inflammation in experimental models of ARDS.

To date, no clinical trial has assessed the effects of early sevoflurane inhalation in ARDS patients.

DESIGN NARRATIVE:

The purpose of this prospective, randomized, controlled study is to evaluate the effects of a 48-hour sevoflurane inhalation strategy on gas exchange and both systemic and pulmonary inflammation in the early phase of ARDS.

After inclusion, ICU patients with moderate to severe ARDS (according to the Berlin definition of ARDS criteria; JAMA 2010) will be randomized into two groups :

* a "conventional group", in which intravenous sedation with midazolam will be administered
* a "sevoflurane group", in which patients will inhale sevoflurane during a 48 hour-period, through dedicated devices Arterial blood gases will be analyze before randomization and at 24, 48, 72, 96, and 120 hours.

Bronchoalveolar lavages (BAL) and blood samples will be assessed before randomization and at 48 hours, in order to measure tumor necrosis factor-alpha (TNFα), interleukin (IL)-1β, IL-6, IL-8 and sRAGE levels. Duplicate assays will be performed with Multiplex (TNFα/interleukins) or ELISA (sRAGE).

During the 48-hour treatment period, bispectral index (BIS®) values ranging from 40 to 50 will be targeted and neuromuscular blocking agents (cisatracurium) will be administered in both groups. Protective ventilation strategies will be applied, as well as other guidelines or recommendations on the management of ICU patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with criteria for moderate to severe ARDS since less than 24 hours (
* Informed consent

Exclusion Criteria:

* Suspected or proven intracranial hypertension
* Midazolam, sevoflurane or cisatracurium allergy
* Medical history of malignant hyperthermia
* Severe liver failure
* Chemotherapy treatment in the last month
* Severe neutropenia (< 0.5 G/l)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | at 48 hours

SECONDARY OUTCOMES:
- Plasma and alveolar levels of proinflammatory cytokines : tumor necrosis factor alpha (TNFα, interleukin (IL)-1β, IL-6, IL-8 | at 48 hours
Plasma and alveolar levels of sRAGE | at 48 hours
PaO2/FiO2 ratio | at day 1, day 3, day 5
Lowest PaO2/FiO2 during the first 5 days of the study | at 5 days
Mean PaO2/FiO2 ratio during the first 5 days of the study | at 5 days
Pulmonary static compliance, resistance and elastance | at day 1, day 2
Duration of controlled mechanical ventilation | at day 30
Total duration of mechanical ventilation (controlled/assisted) | at day 30
Number of ventilatory-free days | at day 30
Number of organ failure-free days | at day 30
Vasopressor requirements | at 48 hours
Mortality | at day 30

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Boucher P, Imhoff E, Chabanne R, Faure JS, Roszyk L, Thibault S, Blondonnet R, Clairefond G, Guerin R, Perbet S, Cayot S, Godet T, Pereira B, Sapin V, Bazin JE, Futier E, Constantin JM. Sevoflurane for Sedation in Acute Respiratory Distress Syndrome. A Randomized Controlled Pilot Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):792-800. doi: 10.1164/rccm.201604-0686OC. PMID 27611637